CLINICAL TRIAL: NCT04546568
Title: Servo Controlled Oxygen Targeting (SCO2T): Servo Versus Servo
Brief Title: SCO2T (Servo vs. Servo)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to meet recruitment target
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AC20034
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2022-05

CONDITIONS: Premature Infant; Oxygen Therapy; Hypoxia; Hyperoxia; Obstetric Labor, Premature
Keywords: Servo Control; Close-Loop Automated Oxygen Control
MeSH Terms: conditions — Premature Birth; Hypoxia; Hyperoxia; Obstetric Labor, Premature

STUDY DESIGN:
Intervention Model Description: This is a randomised cross-over study of servo-controlled oxygen targeting in premature infants, with infants acting as their own controls
Masking Description: This study is randomised but not blinded. Infants will be randomised to commence on either automated (servo) control using either Leoni plus CLAC or IntellO2, Vapotherm. SpO2 (range 90-95%) will be continuously monitored as per normal standard of care.
  To remove selection bias the 20 infants will be randomised using sealed, windowless, envelopes. Half will instruct to commence on automated (servo) control using Leoni plus CLAC (Leoni plus, Löwenstein Medical, Germany) to target SpO2 to 90-95%, and half will have instructions to commence on automated (servo) control using IntellO2 Precision Flow (IntellO2, Vapotherm, USA).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Servo control - Leoni plus CLAC (Experimental): Automated control of oxygen. The oxygen saturation target range will be set to 90-95% as per standard practice.
  Automated oxygen control can be overridden by manual adjustment of oxygen at any time if this is considered necessary to optimise control of oxygenation according to current clinical targets.
  Interventions: Device: Servo control (closed-loop automatic control of the inspiratory fraction of oxygen (FiO2)) - Leoni plus CLAC
- Servo control - IntellO2 Precision Flow, Vapotherm (Active Comparator): Automated control of oxygen. The oxygen saturation target range will be set to 90-95% (set to maintain an integral value of 93%) as per standard practice.
  Automated oxygen control can be overridden by manual adjustment of oxygen at any time if this is considered necessary to optimise control of oxygenation according to current clinical targets.
  Interventions: Device: Servo control (closed-loop automatic control of the inspiratory fraction of oxygen (FiO2)) - IntellO2 OAM

INTERVENTIONS:
Device: Servo control (closed-loop automatic control of the inspiratory fraction of oxygen (FiO2)) - Leoni plus CLAC — FiO2 adjustments will be made by the Leoni plus CLAC (Closed-Loop Automated oxygen Control) ventilator (Leoni plus, Löwenstein Medical, Germany).
  Manual adjustments of the inspired oxygen fraction can additionally be made as per standard care.
  Arms: Servo control - Leoni plus CLAC
Device: Servo control (closed-loop automatic control of the inspiratory fraction of oxygen (FiO2)) - IntellO2 OAM — FiO2 adjustments will be made by the IntellO2 Oxygen Assist Module (OAM) for Precision Flow (IntellO2, Vapotherm, USA).
  Manual adjustments of the inspired oxygen fraction can additionally be made as per standard care.
  Arms: Servo control - IntellO2 Precision Flow, Vapotherm

SUMMARY:
Most premature babies require oxygen therapy. There is uncertainty about what oxygen levels are the best. The oxygen levels in the blood are measured using a monitor called a saturation monitor and the oxygen the baby breathes is adjusted to keep the level in a target range. Although there is evidence that lower oxygen levels maybe harmful, it is not known how high they need to be for maximum benefit. Very high levels are also harmful. Saturation monitors are not very good for checking for high oxygen levels. For this a different kind of monitor, called a transcutaneous monitor, is better.

Keeping oxygen levels stable is usually done by nurses adjusting the oxygen levels by hand (manual control). There is also equipment available that can do this automatically (servo control). It is not known which is best.

Studies of automated control have shown that infants spend more time within their intended target oxygen saturation range. These have not included measurements of transcutaneous oxygen. There are no previous studies directly comparing automated respiratory devices.

The investigators aim to show the transcutaneous oxygen levels as well as the oxygen saturation levels when babies have their oxygen adjusted using two automated (servo) control devices delivering nasal high flow.

For a period of 12 hours each baby will have their oxygen adjusted automatically using each devices for 6 hours respectively. The investigators will compare the range of oxygen levels that are seen between the two respiratory devices.

DETAILED DESCRIPTION:
Presently oxygen is titrated against saturation (SpO2) by manual adjustment. Automated or servo-control systems have been developed that result in tighter control of SpO2 and more time spent in the intended target range. These systems are already in clinical use. Automated systems produce quite large fluctuations in fraction of inspired oxygen (FiO2) in order to keep SpO2 in range. It is possible that this could result in short periods of high or low oxygen tension (PO2) that are undetectable using saturation monitoring. Studies to date have examined the effects of manual and automated (servo) oxygen targeting on SpO2 but not on transcutaneous oxygen tension (TcPO2). There are no studies directly comparing two automated systems.

There is a need to determine the achieved SpO2 and TcPO2 distributions associated with the use of different automated control systems as a first step in planning future trials. When this is measured over a small number of hours it is not anticipated that this would have an influence on clinical outcome.

This study is a prospective, single centre, randomised crossover trial of two automated (servo) control devices - IntellO2 (Vapotherm, USA) versus Leoni plus CLAC (Löwenstein Medical, Germany) - delivering nasal high flow employing automated oxygen titration. Each infant will act as their own control. Infants born at less than 30 weeks gestation, greater than 48 hour of age and receiving supplementary oxygen will be eligible for inclusion.

The study will be undertaken in the Neonatal Unit at the Simpson Centre for Reproductive Health at the Royal Infirmary of Edinburgh.

Total study time is 12 hours for each infant. Infants will be randomised to commence on either automated (servo) control using either Leoni plus CLAC or IntellO2, Vapotherm. SpO2 (range 90-95%) will be continuously monitored as per normal standard of care. A second pulse oximetry probe will be place for servo control input.

Additional monitoring will be carried out as shown below:

1. TcPO2 monitoring
2. FiO2 monitoring
3. Heart rate monitoring (used to validate SpO2 readings)
4. Arterial gas sampling (only if conducted by the direct care team as part of the routine care of the infant; no extra blood samples will be taken as part of the study)

FiO2 will be adjusted by the respiratory support devices which have integrated automated oxygen control, set to maintain a SpO2 target range of 90-95%. The IntellO2 device uses Precision Flow technology (IntellO2, Vapotherm, USA). By means of a modified closed-loop algorithm, the devise uses Masimo pulse oximetry to target a user-set SpO2 value. The Leoni plus CLAC (Closed-Loop Automated oxygen Control) ventilator (Leoni plus, Löwenstein Medical, Germany) similarly uses MasimoSET (Signal Extraction Technology) to target SpO2 and automate oxygen control. Both devices have a signal averaging time of 8 seconds (Masimo, Irvine, USA). The Leoni plus CLAC algorithm is set to a 30 seconds wait time between adjustments, allowing up to 120 automated adjustments/hour.

SpO2 readings will be downloaded directly from the multiparameter patient monitor. SpO2 will be measured using a Phillips MX500 multiparameter monitor (Phillips, Germany, CE 0366). TcPO2 will be measured using a SenTec Digital Monitoring System with OxiVent sensor (SenTec AG, Switzerland, European patent No. 1535055, CE 0120). Both monitors are routinely used in clinical practice. Transcutaneous data will be recorded contemporaneously and the site of the transcutaneous probe will be rotated on each infant every 2 hours. Control of sensor temperature and application duration are designed to meet all applicable standards and this monitoring device is use routinely in many neonatal units.

ELIGIBILITY:
Inclusion Criteria:

1. Infants born at less than 30 weeks gestation
2. Infants greater than 48 hours of age
3. Infants who are receiving supplementary oxygen
4. Person with parental responsibility able to give consent

Exclusion Criteria:

1. Congenital anomalies that would prevent targeting SpO2 to 90-95% (e.g. cardiac defects)
2. Clinical condition of an infant would impair accurateTcPO2 measurement (e.g. impaired perfusion or requirement of inotropic or vasopressor support)

Min Age: 2 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperoxia and hypoxia on transcutaneous monitoring | 12 hours
  To discover the percentage time spent within a TcPO2 range of 50mmHg (6.7kPa) - 80mmHg (10.7kPa) when infants are targeted to an SpO2 range of 90-95% using two automated (servo) control devices (Leoni plus CLAC and Vapotherm IntellO2) delivering nasal high flow.

SECONDARY OUTCOMES:
Transcutanous oxygen variability | 12 hours
  To discover the variability in TcPO2 (measured by standard deviation) when infants are targeted to an SpO2 range of 90-95% using the two automated (servo) control devices delivering nasal high flow.
Incidence of hyperoxia and hypoxia on saturation monitoring | 12 hours
  To discover the percentage time spent within target SpO2 range of 90-95% when infants are targeted using the two automated (servo) control devices delivering nasal high flow.
Saturation variability | 12 hours
  To discover the variability in SpO2 (measured by standard deviation) when infants are targeted to an SpO2 range of 90-95% using the two automated (servo) control devices delivering nasal high flow.
Fraction of inspired oxygen variability | 12 hours
  To discover the variability in FiO2 (measured by standard deviation) when infants are targeted to an SpO2 range of 90-95% using the two automated (servo) control devices delivering nasal high flow.
Pooled frequency histogram of TcPO2 | 12 hours
  To generate a pooled frequency histogram of percentage time at a TcPO2 of below 30mmHg, 30-39.9mmHg, 40-49.9mmHg, 50-59.9mmHg, 60-69.9mmHg, 70-79.9mmHg, and 80mmHg and above for infants targeted to an SpO2 range of 90-95% using the two automated (servo) control devices delivering nasal high flow.
Pooled frequency histogram of SpO2 | 12 hours
  To generate a pooled frequency histogram of percentage time at each SpO2 point between 80 - 100% for infants targeted to an SpO2 range of 90-95% using the two automated (servo) control devices delivering nasal high flow.
Pooled frequency histogram of FiO2 | 12 hours
  To generate a pooled frequency histogram of the cumulative frequency at a FiO2 of 0.21-0.3, 0.31-0.4, 0.41-0.5, 0.51-0.6, 0.61-0.7, 0.81-0.9 and 0.91-1.0 for infants targeted to an SpO2 range of 90-95% using the two automated (servo) control devices delivering nasal high flow.
Desaturations | 12 hours
  To discover the frequency, duration and depth of desaturations and the area (change in PO2 versus time) above and below the set PO2 threshold for infants targeted to an SpO2 range of 90-95% using the two automated (servo) control devices delivering nasal high flow.

CONTACTS AND LOCATIONS:
Locations (1):
- The Simpson Centre for Reproductive Health, Royal Infirmary Edinburgh, Edinburgh, City Of Edinburgh, United Kingdom